CLINICAL TRIAL: NCT07267585
Title: Unravelling the Measles Paradox: a Disease Associated With Both Immune Suppression and Immune Activation
Brief Title: Unravelling the Measles Paradox (MISIA)
Acronym: MISIA
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Corine Geurts van Kessel, Medical microbiologist, Erasmus Medical Center
Other Study IDs: NL-005630
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: MEASLES DISEASE
MeSH Terms: conditions — Measles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample of max 50ml, and give a nasal swab and mucus sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A (receive measles vaccine in 2024): Participant who never had measles vaccine and are recently vaccinated against measles before the upcoming outbreak.
- Group B (not vaccinated, measles infection during upcoming outbreak): Participants who never had measles vaccine and decline recent offer for measles vaccine and get infected with measles during the upcoming outbreak.
- Group C (not vaccinated, no measles infection during upcoming outbreak): Participants who never had measles vaccine and decline recent offer for measles vaccine and remain free from measles infection.
- Group D (not vaccinated, historical infection): Participants who never had measles vaccine and had a history of measles infection.
- Group E (historically vaccinated): Participants who have received measles vaccine about 10 years ago.

SUMMARY:
The measles (MeV) paradox refers to an apparent contradiction: natural measles causes a transient but profound immune suppression putting patients at risk for opportunistic infections for years, while at the same time MeV infection induces robust immune activation leading to lifelong protection against measles. In this protocol, we test our hypothesis that natural measles causes immune amnesia by altering the composition of circulating immune memory cells. In comparison to the prior studies performed during the 2013 outbreak, we will specifically determine [1] to what extent pre-existing immunity is reduced, [2] for how long this functional immune suppression can be detected, and [3] to what extent MeV-specific immune cells expand.

Recently, the WHO reported a 30-fold increase of the number of measles cases in the European Region in 2023 and the ECDC has published a threat assessment brief on increase of the number of cases and considerations for public health response. Combined with the reported drop in vaccination coverage, and several clusters of cases, we anticipate that we are at the verge of a new measles outbreak in the Netherlands

DETAILED DESCRIPTION:
The measles paradox refers to an apparent contradiction: natural measles causes a transient but profound immune suppression putting patients at risk for opportunistic infections for years, while at the same time MeV infection induces robust immune activation leading to lifelong protection against measles. In this protocol, we test our hypothesis that natural measles causes immune amnesia by altering the composition of circulating immune memory cells. In comparison to the prior studies performed during the 2013 outbreak, we will specifically determine [1] to what extent pre-existing immunity is reduced, [2] for how long this functional immune suppression can be detected, and [3] to what extent MeV-specific immune cells expand.

Measles Measles is caused by infection with measles virus (MeV), which is the most contagious human virus known. It is transmitted via aerosols or direct contact with contaminated respiratory secretions and causes systemic disease with clinical signs that appear within two weeks after infection and include fever, rash, cough, coryza and conjunctivitis. Despite significant progress in global measles control programs, every year measles results in the death of more than 100,000 children. Most fatal cases occur in low-income countries, where case-fatality rates often exceed 1% but can be as high as 25% in refugee camps. Case-fatality rates are usually lower than 0.1% in high-income countries; during the Dutch 2013 outbreak, 2,700 cases were reported (real case numbers were likely around 30,000 based on estimated levels of under-reporting), and 1 fatal case was reported in the acute phase of the outbreak. Long-term neurological complications after measles caused two deaths.

Primary infections MeV is often referred to as a respiratory virus, but mainly infects cells of the immune system. Our studies in non-human primates demonstrated how the virus enters the host by infecting alveolar macrophages and dendritic cells in the lungs. After local replication and expansion in the lungs and local lymphoid tissues, MeV disseminated to all peripheral lymphoid tissues. This lymphoid phase was followed by spread to non-lymphoid tissues, including the gingiva, tongue, buccal mucosa, trachea, nose, and skin. Individuals are infectious before the rash appears, and host-to-host transmission is mediated by MeV particles produced by infected epithelial cells in the nose, or MeV-infected lymphocytes in the tonsils and adenoids. Damage to the epithelium of the trachea induces coughing, leading to both cell-free and cell-associated MeV being expelled into the air, which can be inhaled by a next susceptible host. Without complications, patients rapidly recover from measles and are protected for the rest of their life. However, measles transiently suppresses the immune system, leaving patients susceptible to opportunistic infections, like bacterial pneumonia or gastro-intestinal disease.

Lymphopenia and immune amnesia CD150 is the main cellular entry receptor for MeV, which is predominantly present on cells of the immune system. Our previous studies have shown that MeV preferentially infects CD150+ B-cells and central and effector memory T-cells in non-human primates and humans, which are responsible for immunological recall responses. MeV infection and subsequent depletion of B- and memory T-cells explains the measles-induced immune suppression. However, the number of lymphocytes in blood is restored within weeks, so this does not directly explain how immune suppression can last up to years after resolution of measles. We hypothesized that pre-existing immune memory is replaced by measles-specific memory, thus causing immune amnesia. This means that the numbers of antigen-specific lymphocytes are similar before and after measles, but that the repertoire is completely different. This model not only explains the measles paradox, but also why introduction of measles vaccine programs reached further than protection from measles alone.

Functionally, immune amnesia was confirmed by demonstrating disappearance of pre-existing Mantoux responses and impaired responses to prior vaccinations after natural measles. Recently, in vivo studies with canine distemper virus (CDV), a virus closely related to MeV that is used as a model to study immune suppression in ferrets, demonstrated a loss of influenza vaccine responses after CDV infection. Real-world data from African countries showed that the overall disease burden from diarrhoea, lower respiratory infection, malaria, meningitis, and tuberculosis is inversely proportional to measles prevalence. Additionally, the introduction of measles vaccination programs coincided with a drastic decrease in child morbidity and mortality, which could not be explained by the prevention measles alone.

Live attenuated vaccine A safe and effective live-attenuated measles vaccine is available and part of the Dutch national immunization program since 1976. In the Netherlands, the measles vaccine is administered as a trivalent vaccination with mumps and rubella (MMR). The MMR vaccine contains a live attenuated MeV strain that is highly immunogenic in healthy subjects, with measles neutralizing antibodies developing in 90% of individuals after the first dose and 99% after two doses. We have demonstrated in non-human primates that the vaccine virus replicates at a low level in the myeloid cells at the site of injection. It is generally accepted that the measles vaccine does not have an immune suppressive effect and vaccination does not result in lymphopenia, while still inducing lifelong immunity. Given the real-world evidence it is unlikely that the attenuated vaccine strain depletes pre-existing memory cells; yet small changes may go unnoticed as they seem clinically irrelevant. Therefore, subtle changes in the composition of the pre-existing immune repertoire, or the or magnitude of recall responses cannot be excluded.

Duration of measles induced immune suppression In our previous work during the 2013 outbreak, we mainly focused on the short-term effects of natural measles and demonstrated the infection and depletion of circulating immune memory cells. However, post measles blood samples were collected relatively short after recovery. No studies have been conducted yet to fully analyse long-term phenotypical and functional changes in the composition of circulating immune memory cells. Inclusion of controls (vaccinated and uninfected) is crucial for the success of this study.

Trend towards decreasing vaccine uptake and increased measles incidence

In the Dutch national immunization program, the first MMR vaccination is offered at the age of 14 months and the second when the child is 9 years old. Before the introduction of the measles vaccine nearly everyone experienced measles during their childhood, but since the introduction of measles vaccination usually only ±10 cases per year are reported, usually related to import from endemic countries. Although the exact MMR vaccination coverage in the Netherlands cannot be determined by the RIVM because of the implementation of an informed consent for data exchange in January 2022, the current registered percentage of full MMR vaccination is below the 95% needed to prevent transmission chains, and much lower in some regions. The vaccination coverage in the Netherlands shows large regional differences. Vaccine refusal in the Netherlands not only occurs in the Orthodox Protestant community, but also in people with an anthroposophical lifestyle and in certain immigrant populations. Combined, this leads to clusters of low vaccination coverage. For this protocol, we will predominantly (but not exclusively) recruit participants in two communities with low vaccination coverage:

1. The Orthodox Protestant community: The outbreak in 1999-2000 involved 3,381 reported cases and led to 106 hospitalizations, including 3 deaths. The 2012-2013 outbreak involved 2,668 reported cases and 164 hospitalizations, leading to 1 acute and 3 long-term deaths. Since outbreaks occur at an interval of 10-12 years, the time needed to build a large enough group of individuals susceptible to measles, a new outbreak is anticipated.
2. Immigrant population in Rotterdam: Vaccination coverage in Rotterdam is monitored by The Rotterdam Outbreak Surveillance Team' (ROST), a collaboration between the Erasmus MC department of Viroscience, the GGD Rotterdam, and the Erasmus MC Pandemic and Disaster Preparedness Center. Coverage of the two-dose vaccination schedule in Rotterdam is estimated at 76%; however, in some neighbourhoods and schools it has apparently dropped below 45%. Outbreaks in these clusters of low vaccination coverage are a realistic possibility.

On the verge of an outbreak Recently, the WHO reported a 30-fold increase of the number of measles cases in the European Region in 2023 and the ECDC has published a threat assessment brief on increase of the number of cases and considerations for public health response. Combined with the reported drop in vaccination coverage, and several clusters of cases, we anticipate that we are at the verge of a new measles outbreak in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

Cohort A

* 18 years or older
* No known history of measles or vaccination
* Decided to take MMR vaccination before the upcoming measles outbreak

Cohort B

* 18 years or older
* No known history of measles or vaccination (seronegative confirmed)
* Contracted measles during the upcoming outbreak

Cohort C

* 18 years or older
* No known history of measles or vaccination (seronegative confirmed)

Cohort D

* 18 years or older
* Experienced measles during the 2013 outbreak

Cohort E

* 18 years or older
* Received second dose of measles vaccines ±10 years ago

Exclusion Criteria:

A potential participant who meets any of the following criteria will be excluded from the study:

* Diagnosed chronic disease
* Immune suppression (due to medication or underlying disease)
* Additionally for subjects recruited to Cohort A:

  * pregnant women or women planning to get pregnant in less than one month after the start of the study. This is a precaution; the MMR vaccine is not recommended for pregnant women.
  * People who have had a severe allergic reaction (e.g., anaphylaxis) after a previous vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants in this study are 18 years or older and will be recruited in areas with low vaccination coverage. Recruitment will occur through contacting orthodox protestant student associations, GPs with a large orthodox protestant patient base, orthodox protestant newspapers, and first year medical students at the Erasmus MC. The study does not include an intervention.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Compare measles-induced loss of pathogen-specific antibodies | 36 months
  The investigators will measure changes in the immune repertoire using longitudinal samples obtained from participants who are infected with MeV. To this end, they will measure pathogen-specific antibody responses (titers) pre- and post-measles and compare these to determine whether measles led to a loss of pathogen-specific antibodies.
Compare measles-induced loss of pathogen-specific T-cells | 36 months
  The investigators will measure changes in the immune repertoire using longitudinal samples obtained from participants who are infected with MeV. To this end, they will measure pathogen-specific T-cell responses (frequencies) pre- and post-measles and compare these to determine whether measles led to a loss of pathogen-specific T-cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Knol M, Urbanus A, Swart E, Mollema L, Ruijs W, van Binnendijk R, Te Wierik M, de Melker H, Timen A, Hahne S. Large ongoing measles outbreak in a religious community in the Netherlands since May 2013. Euro Surveill. 2013 Sep 5;18(36):pii=20580. doi: 10.2807/1560-7917.es2013.18.36.20580. PMID 24079377
- [Background] Van Den Hof S, Smit C, Van Steenbergen JE, De Melker HE. Hospitalizations during a measles epidemic in the Netherlands, 1999 to 2000. Pediatr Infect Dis J. 2002 Dec;21(12):1146-50. doi: 10.1097/00006454-200212000-00012. PMID 12488666
- [Background] van Velzen E, de Coster E, van Binnendijk R, Hahne S. Measles outbreak in an anthroposophic community in The Hague, The Netherlands, June-July 2008. Euro Surveill. 2008 Jul 31;13(31):18945. No abstract available. PMID 18761905
- [Background] Mollema L, Harmsen IA, Broekhuizen E, Clijnk R, De Melker H, Paulussen T, Kok G, Ruiter R, Das E. Disease detection or public opinion reflection? Content analysis of tweets, other social media, and online newspapers during the measles outbreak in The Netherlands in 2013. J Med Internet Res. 2015 May 26;17(5):e128. doi: 10.2196/jmir.3863. PMID 26013683
- [Background] Laksono BM, de Vries RD, Verburgh RJ, Visser EG, de Jong A, Fraaij PLA, Ruijs WLM, Nieuwenhuijse DF, van den Ham HJ, Koopmans MPG, van Zelm MC, Osterhaus ADME, de Swart RL. Studies into the mechanism of measles-associated immune suppression during a measles outbreak in the Netherlands. Nat Commun. 2018 Nov 23;9(1):4944. doi: 10.1038/s41467-018-07515-0. PMID 30470742
- [Background] Mina MJ, Kula T, Leng Y, Li M, de Vries RD, Knip M, Siljander H, Rewers M, Choy DF, Wilson MS, Larman HB, Nelson AN, Griffin DE, de Swart RL, Elledge SJ. Measles virus infection diminishes preexisting antibodies that offer protection from other pathogens. Science. 2019 Nov 1;366(6465):599-606. doi: 10.1126/science.aay6485. PMID 31672891
- [Background] Rennick LJ, de Vries RD, Carsillo TJ, Lemon K, van Amerongen G, Ludlow M, Nguyen DT, Yuksel S, Verburgh RJ, Haddock P, McQuaid S, Duprex WP, de Swart RL. Live-attenuated measles virus vaccine targets dendritic cells and macrophages in muscle of nonhuman primates. J Virol. 2015 Feb;89(4):2192-200. doi: 10.1128/JVI.02924-14. Epub 2014 Dec 3. PMID 25473055
- [Background] de Vries RD, Lemon K, Ludlow M, McQuaid S, Yuksel S, van Amerongen G, Rennick LJ, Rima BK, Osterhaus AD, de Swart RL, Duprex WP. In vivo tropism of attenuated and pathogenic measles virus expressing green fluorescent protein in macaques. J Virol. 2010 May;84(9):4714-24. doi: 10.1128/JVI.02633-09. Epub 2010 Feb 24. PMID 20181691
- [Background] Aaby P, Bukh J, Lisse IM, Smits AJ. Measles vaccination and reduction in child mortality: a community study from Guinea-Bissau. J Infect. 1984 Jan;8(1):13-21. doi: 10.1016/s0163-4453(84)93192-x. PMID 6699411
- [Background] Sato R, Haraguchi M. Effect of measles prevalence and vaccination coverage on other disease burden: evidence of measles immune amnesia in 46 African countries. Hum Vaccin Immunother. 2021 Dec 2;17(12):5361-5366. doi: 10.1080/21645515.2021.2013078. Epub 2021 Dec 29. PMID 34965183
- [Background] Petrova VN, Sawatsky B, Han AX, Laksono BM, Walz L, Parker E, Pieper K, Anderson CA, de Vries RD, Lanzavecchia A, Kellam P, von Messling V, de Swart RL, Russell CA. Incomplete genetic reconstitution of B cell pools contributes to prolonged immunosuppression after measles. Sci Immunol. 2019 Nov 1;4(41):eaay6125. doi: 10.1126/sciimmunol.aay6125. PMID 31672862
- [Background] Cox RM, Wolf JD, Lieberman NA, Lieber CM, Kang HJ, Sticher ZM, Yoon JJ, Andrews MK, Govindarajan M, Krueger RE, Sobolik EB, Natchus MG, Gewirtz AT, deSwart RL, Kolykhalov AA, Hekmatyar K, Sakamoto K, Greninger AL, Plemper RK. Therapeutic mitigation of measles-like immune amnesia and exacerbated disease after prior respiratory virus infections in ferrets. Nat Commun. 2024 Feb 8;15(1):1189. doi: 10.1038/s41467-024-45418-5. PMID 38331906
- [Background] Laksono BM, Roelofs D, Comvalius AD, Schmitz KS, Rijsbergen LC, Geers D, Nambulli S, van Run P, Duprex WP, van den Brand JMA, de Vries RD, de Swart RL. Infection of ferrets with wild type-based recombinant canine distemper virus overwhelms the immune system and causes fatal systemic disease. mSphere. 2023 Aug 24;8(4):e0008223. doi: 10.1128/msphere.00082-23. Epub 2023 Jun 28. PMID 37377421
- [Background] Ward BJ, Johnson RT, Vaisberg A, Jauregui E, Griffin DE. Cytokine production in vitro and the lymphoproliferative defect of natural measles virus infection. Clin Immunol Immunopathol. 1991 Nov;61(2 Pt 1):236-48. doi: 10.1016/s0090-1229(05)80027-3. PMID 1914259
- [Background] Hirsch RL, Griffin DE, Johnson RT, Cooper SJ, Lindo de Soriano I, Roedenbeck S, Vaisberg A. Cellular immune responses during complicated and uncomplicated measles virus infections of man. Clin Immunol Immunopathol. 1984 Apr;31(1):1-12. doi: 10.1016/0090-1229(84)90184-3. PMID 6230187
- [Background] Tamashiro VG, Perez HH, Griffin DE. Prospective study of the magnitude and duration of changes in tuberculin reactivity during uncomplicated and complicated measles. Pediatr Infect Dis J. 1987 May;6(5):451-4. doi: 10.1097/00006454-198705000-00007. PMID 3601492
- [Background] de Vries RD, McQuaid S, van Amerongen G, Yuksel S, Verburgh RJ, Osterhaus AD, Duprex WP, de Swart RL. Measles immune suppression: lessons from the macaque model. PLoS Pathog. 2012;8(8):e1002885. doi: 10.1371/journal.ppat.1002885. Epub 2012 Aug 30. PMID 22952446
- [Background] de Swart RL, Ludlow M, de Witte L, Yanagi Y, van Amerongen G, McQuaid S, Yuksel S, Geijtenbeek TB, Duprex WP, Osterhaus AD. Predominant infection of CD150+ lymphocytes and dendritic cells during measles virus infection of macaques. PLoS Pathog. 2007 Nov;3(11):e178. doi: 10.1371/journal.ppat.0030178. PMID 18020706
- [Background] Mina MJ, Metcalf CJ, de Swart RL, Osterhaus AD, Grenfell BT. Long-term measles-induced immunomodulation increases overall childhood infectious disease mortality. Science. 2015 May 8;348(6235):694-9. doi: 10.1126/science.aaa3662. Epub 2015 May 7. PMID 25954009
- [Background] Ludlow M, Lemon K, de Vries RD, McQuaid S, Millar EL, van Amerongen G, Yuksel S, Verburgh RJ, Osterhaus AD, de Swart RL, Duprex WP. Measles virus infection of epithelial cells in the macaque upper respiratory tract is mediated by subepithelial immune cells. J Virol. 2013 Apr;87(7):4033-42. doi: 10.1128/JVI.03258-12. Epub 2013 Jan 30. PMID 23365435
- [Background] Ludlow M, de Vries RD, Lemon K, McQuaid S, Millar E, van Amerongen G, Yuksel S, Verburgh RJ, Osterhaus ADME, de Swart RL, Duprex WP. Infection of lymphoid tissues in the macaque upper respiratory tract contributes to the emergence of transmissible measles virus. J Gen Virol. 2013 Sep;94(Pt 9):1933-1944. doi: 10.1099/vir.0.054650-0. Epub 2013 Jun 19. PMID 23784446
- [Background] Lemon K, de Vries RD, Mesman AW, McQuaid S, van Amerongen G, Yuksel S, Ludlow M, Rennick LJ, Kuiken T, Rima BK, Geijtenbeek TB, Osterhaus AD, Duprex WP, de Swart RL. Early target cells of measles virus after aerosol infection of non-human primates. PLoS Pathog. 2011 Jan 27;7(1):e1001263. doi: 10.1371/journal.ppat.1001263. PMID 21304593
- [Background] Laksono BM, de Vries RD, McQuaid S, Duprex WP, de Swart RL. Measles Virus Host Invasion and Pathogenesis. Viruses. 2016 Jul 28;8(8):210. doi: 10.3390/v8080210. PMID 27483301
- [Background] Laksono BM, de Vries RD, Duprex WP, de Swart RL. Measles pathogenesis, immune suppression and animal models. Curr Opin Virol. 2020 Apr;41:31-37. doi: 10.1016/j.coviro.2020.03.002. Epub 2020 Apr 24. PMID 32339942
- [Background] de Vries RD, de Swart RL. Measles immune suppression: functional impairment or numbers game? PLoS Pathog. 2014 Dec 18;10(12):e1004482. doi: 10.1371/journal.ppat.1004482. eCollection 2014 Dec. No abstract available. PMID 25522010
- See also: WHO measles key facts — https://www.who.int/news-room/fact-sheets/detail/measles?gclid=Cj0KCQjwuZGnBhD1ARIsACxbAVhFlwf3glmjE80pXyz9hyY00pt0ZIpT8OzPDelzCVua5776SP8iZMsaAjqbEALw_wcB
- See also: A 30-fold rise of measles cases in 2023 in the WHO European Region warrants urgent action — https://www.who.int/europe/news/item/14-12-2023-a-30-fold-rise-of-measles-cases-in-2023-in-the-who-european-region-warrants-urgent-action
- See also: Measles on the rise in the EU/EEA: considerations for public health response — https://www.ecdc.europa.eu/sites/default/files/documents/measles-eu-threat-assessment-brief-february-2024.pdf